CLINICAL TRIAL: NCT04451174
Title: Early Use of Corticosteroids in Non-critical Patients With COVID-19 Pneumonia (PREDCOVID)
Brief Title: Early Use of Corticosteroids in Non-critical Patients With COVID-19 Pneumonia
Acronym: PREDCOVID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Corticosteroid use approval
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Mauricio Salinas, Mauricio Salinas MD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2092
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Prednisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Prednisone 40 mg days 1 to 4. Then Prednisone 20 mg days 5 to 8.
  Interventions: Drug: Prednisone
- Control (No Intervention)

INTERVENTIONS:
Drug: Prednisone — Prednisone 40 mg days 1 to 4. Then, prednisone 20 mg days 5 to 8.
  Arms: Treatment

SUMMARY:
Steroids has shown benefits in COVID19 patients in observational studies. We hypothesized that early use of corticosteroids, low dose, in mild disease, can decrease progression to respiratory failure and death.

DETAILED DESCRIPTION:
We are in the middle of a coronavirus pandemic, facing a large number of infections in serious cases and an increasing number of deaths in Chile. As of June 11, 2020, there are 154092 cases confirmed by COVID - 19 i and 2648 deaths in our country.

Most patients have mild disease, but older people and those with comorbidities can develop severe disease that requires hospitalization, some form of ventilatory support, and eventually intensive care unit admission. The pathophysiology occurs in two different overlapping phases, the initial pathogen with viral replication, followed by the host's inflammatory response with varying degrees of severity associated with different clinical characteristics. The pathological progression in some cases of severe COVID-19 would be explained by an excess of proinflammatory cytokines, which leads to diffuse alveolar damage, with the development of acute respiratory distress syndrome (ARDS) and inflammatory compromise of multiple systems until death.

In the absence of any proven antiviral therapy, current clinical treatment is primarily supportive care, supplemental oxygen, and mechanical ventilatory support.

Clinical trials have been published and called to demonstrate the usefulness of therapies in the context of this pandemic.

The role of corticosteroids is not fully defined. Observational studies report better results in decreasing disease progression in those COVID-19 patients who received corticosteroids early.

We hypothesize in this study that treatment in mild disease (defined as that requiring supplemental oxygen, but without the need for ventilatory support) can attenuate the host's excessive respiratory and systemic inflammatory responses.

The objective of this study is to evaluate the effect of early treatment with prednisone to decrease the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* COVID-19 confirmed by PCR
* Oxygen requirements until 35 % by venturi mask or 5 lt minutes by nasal cannula
* Consent form signed

Exclusion Criteria:

* Previous steroid use 48 hours or more.
* Pregnancy
* Chronic respiratory failure
* Requirements of mechanical ventilation (invasive or no invasive)
* Chronic liver damage Child Pugh B or C
* Chronic kidney disease stage IV or V.
* Immunosuppressed
* Participation on other trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Composite Primary End-point: Admission to ICU, Need for Invasive Mechanical Ventilation or All-cause Death by Day 28 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Salinas, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Santiago Oriente, Santiago, Peñalolen, Chile

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication

REFERENCES:
- [Derived] Salinas M, Andino P, Palma L, Valencia J, Figueroa E, Ortega J. Early use of corticosteroids in non-critical patients with COVID-19 pneumonia (PREDCOVID): a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Jan 26;22(1):92. doi: 10.1186/s13063-021-05046-6. PMID 33499887